CLINICAL TRIAL: NCT07275242
Title: An Open-Label, Multi-site Phase I Clinical Study of SHR-A1811(sc) Subcutaneous Injection: Evaluating Pharmacokinetics, Safety, Tolerability, and Efficacy in Patients With Solid Tumor
Brief Title: A Clinical Study of SHR-A1811(sc) Subcutaneous Injection in Patients With Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811(sc)-101
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose Group (Experimental)
  Interventions: Drug: SHR-A1811 Subcutaneous Injection; Drug: SHR-A1811 for Injection
- Medium-Dose Group (Experimental)
  Interventions: Drug: SHR-A1811 Subcutaneous Injection; Drug: SHR-A1811 for Injection
- High-Dose Group (Experimental)
  Interventions: Drug: SHR-A1811 Subcutaneous Injection; Drug: SHR-A1811 for Injection

INTERVENTIONS:
Drug: SHR-A1811 Subcutaneous Injection — SHR-A1811 subcutaneous injection.
Drug: SHR-A1811 for Injection — SHR-A1811 for injection.

SUMMARY:
The study is being conducted to evaluate the pharmacokinetics , safety, tolerability and efficacy in patients with solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. Solid Tumor confirmed by histology or cytology;
3. ECOG score is 0 or 1;
4. An expected survival of ≥ 12 weeks;
5. At least one measurable lesion according to RECIST v1.1 criteria;
6. Have adequate renal and hepatic function;
7. Patients voluntarily joined the study and signed informed consent.

Exclusion Criteria:

1. With a history of any malignancies in the past 5 years, excluding cured cervical carcinoma in situ and melanoma skin cancer;
2. Patients have major surgical procedures or radiotherapy / chemotherapy within 4 weeks before the first medication;
3. History of immunodeficiency;
4. Clinically significant cardiovascular diseases;
5. Known or suspected interstitial lung disease;
6. Known hereditary or acquired bleeding thrombotic tendency;
7. Active hepatitis and liver cirrhosis;
8. Known allergic history of the drug components of this protocol;
9. History of neurological or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to 21 days (AUC0-21d) of SHR-A1811(sc) | About 72 weeks.
The incidence and severity of Dose-Limiting Toxicities (DLTs) | About 72 weeks.
Adverse Events (AEs) | About 72 weeks.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | About 72 weeks.
Maximum concentration (Cmax) | About 72 weeks.
Trough concentration (Cmin) | About 72 weeks.
Area under the concentration-time curve from time zero to the time of the last measurable concentration (AUC0-t) | About 72 weeks.
Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) | About 72 weeks.
Elimination half-life (t1/2) | About 72 weeks.
Mean residence time (MRT) | About 72 weeks.
Apparent clearance (CL/F) | About 72 weeks.
Apparent volume of distribution at steady state (Vss/F) | About 72 weeks.
Area under the concentration-time curve at steady state (AUCss) | About 72 weeks.
Maximum concentration at steady state (Css, max) | About 72 weeks.
Trough concentration at steady state (Css, min) | About 72 weeks.
Accumulation ratio (Rac) | About 72 weeks.
Anti-SHR-A1811 antibodies (ADA) | About 72 weeks.
Objective Response Rate (ORR) | About 72 weeks.
Duration of Response (DoR) | About 72 weeks.
Disease Control Rate (DCR) | About 72 weeks.
Progression-Free Survival (PFS) | About 72 weeks.
Overall Survival (OS) | About 72 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided